CLINICAL TRIAL: NCT01493154
Title: A Phase I Clinical Trial Assessing the Safety and Feasibility of Administration of pNGVL4a-CRT/E7(Detox) DNA Vaccine Using the Intramuscular TriGridTM Delivery System in Combination With Cyclophosphamide in HPV-16 Associated Head and Neck Cancer Patients
Brief Title: Safety Study of HPV DNA Vaccine to Treat Head and Neck Cancer Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study Funding Terminated
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH); Ichor Medical Systems Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J11129; P50DE019032 (NIH); NA_00023916 (Other: JHMIRB)
Record Dates: First submitted 2011-11-21; First posted 2011-12-15 (Estimated); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Head and Neck Cancer
Keywords: HPV; Head and Neck Cancer; Vaccine; Immunotherapy; Cyclophosphamide; Sexually Transmitted Diseases, Viral
MeSH Terms: conditions — Head and Neck Neoplasms; Sexually Transmitted Diseases, Viral | interventions — Vaccines, DNA; detox adjuvant; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cohort 1 - DNA Vaccine (Dose 0.5 mg/dose) (Experimental): pNGVL-4a-CRT/E7 (detox) DNA Vaccine (Dose 0.5 mg/dose) + Cyclophosphamide (200 mg/m2)
  Interventions: Biological: DNA Vaccine; Drug: Cyclophosphamide
- Cohort 2 - DNA Vaccine (Dose 1.0 mg/dose) (Experimental): pNGVL-4a-CRT/E7 (detox) DNA Vaccine (Dose 1.0 mg/dose) + Cyclophosphamide (200 mg/m2)
  Interventions: Biological: DNA Vaccine; Drug: Cyclophosphamide
- Cohort 3 - DNA Vaccine (Dose 2.0 mg/dose) (Experimental): pNGVL-4a-CRT/E7 (detox) DNA Vaccine (Dose 2.0 mg/dose) + Cyclophosphamide (200 mg/m2)
  Interventions: Biological: DNA Vaccine; Drug: Cyclophosphamide
- Cohort 4 - DNA Vaccine (Dose 4.0 mg/dose) (Experimental): pNGVL-4a-CRT/E7 (detox) DNA Vaccine (Dose 4.0 mg/dose) + Cyclophosphamide (200 mg/m2)
  Interventions: Biological: DNA Vaccine; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: DNA Vaccine — Patients will receive intramuscular needle injections of pNGVL4a-CRT/E7 (detox) DNA vaccine using the TDS-IM device on Day 1, 22, and 43 for a total of three vaccinations per patient. One day prior to each DNA vaccination, the patient will receive a single low dose of 200 mg/m2 of cyclophosphamide intravenously. The DNA vaccine will be administered in a dose-escalating manner.
  Other Names: pNGVL-4a-CRT/E7 (detox) DNA Vaccine
Drug: Cyclophosphamide — A single low dose of 200 mg/m2 of cyclophosphamide (CTX) will be administered intravenously up to 24 hours (Day 0) prior to each DNA vaccination.
  Other Names: Cytoxan

SUMMARY:
This study will test the safety of an HPV DNA vaccine after it is injected into your muscle using an electroporation device (TriGridTM Delivery System made by Ichor Medical Systems), and will test the ability of the vaccine to help your body's immune system to recognize HPV-infected and associated cancer cells. In addition to giving the vaccine using an electroporation device, we are giving the vaccine in combination with an immunomodulatory agent to further enhance immune responses against HPV-infected and associated cancer cells.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed diagnosis of squamous cell carcinoma of the head and neck or unknown primary with level II/III (jugulodigastric) nodal involvement (which have been found in previous studies to be the result of subclinical oropharyngeal carcinoma).
2. Head and neck cancer patients documented to have HPV-16 DNA within their tumors as determined by in situ hybridization are eligible for this study.
3. Fresh-frozen or paraffin-embedded material must be available for in situ hybridization testing for HPV-16 DNA.
4. Staging criteria established by the American Joint Committee on Clinical Investigation (AJCC, Fifth Edition, 1997) for Stage III (T1-3N1M0, T3N0M0) or IV (T1-4N2M0, T4N0-1M0 ) disease.
5. Age ≥ 18 years
6. Life expectancy of greater than 4 months.
7. Baseline Eastern Cooperative Oncology Group performance status of 0, 1 at the time of multi-modality treatment administration.

9. Patients must have adequate organ function at the time of enrollment as defined by the following parameters: white blood cell count > 3,000 lymphocyte number > 500 absolute neutrophil count > 1,000 platelets > 90,000 hemoglobulin > 9 total bilirubin <3 X the institutional limit of normal AST(SGOT)/ALT(SGPT) <3 X the institutional limit of normal creatinine < 2.5X the institutional limit of normal

Exclusion Criteria:

1. Diagnosis of immunosuppression or prolonged, active use of immunosuppressive medications such as steroids.
2. Prior enrollment in any vaccine study in the past 24 months.
3. Presence of uncontrolled concurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with study requirements.
4. Presence or history of autoimmune disease such as multiple sclerosis, exclusive of a history of thyroiditis, psoriasis, inflammatory bowel disease, or Sjogren's syndrome.
5. Pregnancy or breast feeding. Pregnancy is defined as any female subject of reproductive potential [defined as girls who have reached menarche or women who have not been post-menopausal for at least 24 consecutive months, i.e., who have had menses within the preceding 24 months, or have not undergone surgical sterilization (e.g., hysterectomy, bilateral oophorectomy, or bilateral tubal ligation)] must have a negative serum -hcg test within 3 days prior to study entry.
6. History of prior malignancy permitted if patient has been disease free for ≥ 5 years, however individuals with completely resected basal cell or squamous cell carcinoma of the skin within this interval may be enrolled.
7. Inability to understand or unwillingness to sign an informed consent document.
8. Patients with a history of arterial or venous thrombosis.
9. Patients with non-healed wounds.
10. Patients with chronic infection with or a history of Hepatitis B, Hepatitis C, or HIV infection as determined by serology tests obtained during the eligibility screening.
11. Current use of any electronic stimulation device, such as cardiac demand pacemakers, automatic implantable cardiac defibrillator, nerve stimulators, or deep brain stimulators.
12. History of, or documented in an EKG within 30 days of study eligibility screening, cardiac arrhythmia or palpitations [e.g., supraventricular tachycardia, atrial fibrillation, frequent ectopy, or sinus bradycardia (i.e., <50 beats per minute on exam)] prior to study entry.

    NOTE: Sinus arrhythmia is not excluded.
13. History of syncope or fainting episode within 1 year of study entry.
14. Seizure disorder or any history of prior seizure.
15. Presence of any surgical or traumatic metal implants at the site of administration (deltoid muscles).
16. Bleeding disorder or other contraindication for intramuscular injection.
17. A skin-fold measurement of the cutaneous and subcutaneous tissue that exceeds 40mm at one or more of the eligible injection sites (the medial deltoid muscles).
18. History of axillary lymph node dissection.
19. Patients who have had chemotherapy or radiotherapy within 28 days (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 28 days earlier.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-04; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events after administration of pNGVL4a-CRT/E7 (detox) DNA vaccine using the intramuscular TriGridTM Delivery System (TDS-IM) in combination with cyclophosphamide | 5 years

SECONDARY OUTCOMES:
Number of participants with measurable HPV-specific immune responses after vaccination | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Califano, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center, Johns Hopkins Hospital
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center, Johns Hopkins Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Background] Cheng WF, Hung CF, Chai CY, Hsu KF, He L, Ling M, Wu TC. Tumor-specific immunity and antiangiogenesis generated by a DNA vaccine encoding calreticulin linked to a tumor antigen. J Clin Invest. 2001 Sep;108(5):669-78. doi: 10.1172/JCI12346. PMID 11544272
- [Background] Best SR, Peng S, Juang CM, Hung CF, Hannaman D, Saunders JR, Wu TC, Pai SI. Administration of HPV DNA vaccine via electroporation elicits the strongest CD8+ T cell immune responses compared to intramuscular injection and intradermal gene gun delivery. Vaccine. 2009 Sep 4;27(40):5450-9. doi: 10.1016/j.vaccine.2009.07.005. Epub 2009 Jul 19. PMID 19622402
- [Background] Vasan S, Hurley A, Schlesinger SJ, Hannaman D, Gardiner DF, Dugin DP, Boente-Carrera M, Vittorino R, Caskey M, Andersen J, Huang Y, Cox JH, Tarragona-Fiol T, Gill DK, Cheeseman H, Clark L, Dally L, Smith C, Schmidt C, Park HH, Kopycinski JT, Gilmour J, Fast P, Bernard R, Ho DD. In vivo electroporation enhances the immunogenicity of an HIV-1 DNA vaccine candidate in healthy volunteers. PLoS One. 2011;6(5):e19252. doi: 10.1371/journal.pone.0019252. Epub 2011 May 16. PMID 21603651
- [Background] Emens LA, Asquith JM, Leatherman JM, Kobrin BJ, Petrik S, Laiko M, Levi J, Daphtary MM, Biedrzycki B, Wolff AC, Stearns V, Disis ML, Ye X, Piantadosi S, Fetting JH, Davidson NE, Jaffee EM. Timed sequential treatment with cyclophosphamide, doxorubicin, and an allogeneic granulocyte-macrophage colony-stimulating factor-secreting breast tumor vaccine: a chemotherapy dose-ranging factorial study of safety and immune activation. J Clin Oncol. 2009 Dec 10;27(35):5911-8. doi: 10.1200/JCO.2009.23.3494. Epub 2009 Oct 5. PMID 19805669
- See also: Related Info — http://www.hopkinsmedicine.org/kimmel_cancer_center/centers/head_neck/research_studies_and_clinical_trials/